CLINICAL TRIAL: NCT02450955
Title: Does the Addition of Manipulation Provide Added Benefit to Massage Therapy for Tension-type Headache Patients? A Randomized Controlled Clinical Trial
Brief Title: Does the Addition of Manipulation Provide Added Benefit to Massage Therapy for Tension-type Headache Patients?
Acronym: MANIHDI-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, PhD, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ID006
Record Dates: First submitted 2015-05-17; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Tension-type Headache
Keywords: Tension-type headache; manual therapy; disability; spinal manipulation
MeSH Terms: conditions — Tension-Type Headache | interventions — Massage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Massage (Active Comparator): A superficial massage was performed for 10 minutes in the cervical region consisting of gentle rubbing and kneading.
  Interventions: Other: Massage
- Occiput-Atlas-Axis Technique (Experimental): The technique is applied in two stages: in the first stage, a light core decompression is performed and then small circumductions are made with the aim of increasing viscoelasticity of tissues. Subsequently the appropriate joint barrier is sought by selective tension and high-velocity rotation manipulation is performed in a cranial helical motion without raising the subjects head.
  Interventions: Other: Occiput-Atlas-Axis Technique

INTERVENTIONS:
Other: Massage — A superficial massage was performed for 10 minutes in the cervical region consisting of gentle rubbing and kneading, five minutes prone and five minutes supine with a focus on cervical and suboccipital muscles in order to induce a global relaxation of the cervical and suboccipital region. Resting position. After the treatment, both groups rested for 10 minutes in a supine position with neutral ranges of neck flexion, extension, lateral flexion, and rotation.
  Other Names: Active Comparator
  Arms: Massage
Other: Occiput-Atlas-Axis Technique — This technique was applied as described previously and is used with the aim of restoring joint mobility between the occiput, atlas and axis. It is a structural technique applied bilaterally, performed on a vertical axis passing through the dens process of the axis without extension or flexion and very little side-bending. After the treatment, both groups rested for 10 minutes in a supine position with neutral ranges of neck flexion, extension, lateral flexion, and rotation.
  Other Names: Experimental
  Arms: Occiput-Atlas-Axis Technique

SUMMARY:
Objective. To compare the benefits of spinal manipulation combined with massage therapy versus massage alone in patients with tension-type headache (TTH) on the frequency, intensity and disability caused by headache and on cervical range of motion.

Method. A factorial, randomized, double-blinded, placebo-controlled clinical trial was conducted with a sample of 105 subjects diagnosed with TTH, divided into two groups: a) the treatment group received a manipulative technique followed by massage of the cervical and suboccipital region; a) the control group received massage alone. Four sessions (once per week) were applied over four weeks. The Headache Disability Inventory (HDI) was used to evaluate changes in the frequency and severity of headache and functional and emotional aspects of headache. Range of upper cervical and cervical flexion and extension were evaluated. Measures were conducted at baseline, immediately after the intervention (week 4) and at a follow up 8 weeks after completion of the intervention.

DETAILED DESCRIPTION:
MATERIALS AND METHODS Participants The sample consisted of 105 people diagnosed with frequent (47.6%) and chronic (52.4%) TTH derived from two primary care centres, selected according to the criteria of IHS3,4, and suffering from headache for more than three months. Participants were aged between 18 and 65 years (mean ± SD: 38.9 ± 10.9 years), which included 23 men (21.9%) and 82 women (78.1%). Patients were excluded if they had suspected malignant disease, rheumatoid arthritis, pregnancy, vertigo, continuous intake of prescribed medication or those who received physical therapy in the past 3 months for headache or neck pain. Finally, 102 subjects completed the study (2 from the treatment group dropped out due to work problems and one from the control due to lack of improvement).

The software G*power14 was to calculate the required sample size, using data from previous studies to estimate the effect sizes to be expected. Our review of the extant literature showed that across studies, the mean N was 44.28 and in general large effect sizes were found (Cohen's d = .40).15-19 We accepted a 5% alpha risk (α = .05) and 10% beta risk (β = .1) as study parameters which showed that 51 subjects were required in each group to achieve a medium-to-large effect size (f = .35). We predicted a 5% dropout rate in the follow-up period.

Study design The study was a factorial, randomized, double-blinded, placebo-controlled clinical trial. It was conducted from January to November, 2014. After the initial clinical interview, the allocation of patients to control or treatment groups was randomized by an external assistant using a specific software (name) who monitored the sequence and documentation at all times. Both the external assistant and the therapist and examiner were blinded to the study objective.

Patients were randomly assigned into 2 groups (treatment and control). The treatment group received occiput-atlas-axis manipulation (OAA) and soft tissue treatment by massage. The control group received massage only. Thus both groups received the same duration of massage therapy and the exposure times were the same, however the difference between groups lay in the manipulative OAA technique which only the treatment group received. Four sessions were conducted (once per week) and the assessment was carried out in 3 stages: at baseline, end of treatment (at 4 weeks) and follow-up at 8 weeks following completion of treatment. All patients in both groups were assessed under the same conditions before and after the treatment by an examiner blinded to the group allocation.

The study was conducted at the University of Valencia (Spain) from January 2014 to November 2014. Prior to data collection, informed written consent was obtained from all patients, and all procedures were conducted according to the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 65 years
* Diagnosis of frequent ETTH and CTTH
* Having headache episodes on more than 4 days per month
* Headache episodes lasting from 30 minutes to 7 days
* Headaches having at least 2 of the following characteristics:

  * Bilateral location of pain
  * Pressing non pulsating quality
  * Mild or moderate intensity
  * Not aggravated by physical activity
* Sufferers may present photophobia, phonophobia, nausea or vomiting
* Headache may be associated with pericranial tenderness
* Suffering from TTH for over 3 months
* Subjects being under pharmacological control

Exclusion Criteria:

* • Patients with infrequent ETTH, and patients with probable TTH in its frequent and infrequent forms.

  * Headache that is aggravated by head movements.
  * Metabolic or musculoskeletal disorders with symptoms similar to headache (rheumatoid arthritis)
  * Previous neck trauma
  * Vertigo, dizziness, arterial hypertension.
  * Joint stiffness, arteriosclerosis or advanced degenerative osteoarthritis
  * Patients with heart devices
  * Patients in process of pharmacological adaptation
  * Excessive emotional tension
  * Neurological disorders
  * Laxity of neck soft tissues
  * Radiological alterations
  * General hypermobility or hyperlaxity
  * Joint instability
  * Pregnancy
  * Received physical therapy treatment for headache or neck pain in the previous 3 months
  * Suspicion of malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Headache Disability Inventory (HDI). | 8 weeks
  An inventory of disability caused by headaches developed by Jacobson et al. and Gary et al. was used. The purpose of the scale is to identify the difficulties the patient may experience due to headache. It includes 2 items: headache severity (mild, moderate and severe) and frequency (once a month, more than once and less than 4 times a month, and once a week) and 25 items that assess two subscales (E = Emotional with 13 items and F = Functional, with 12 items). Subjects answer each question (yes = 4 points, sometimes = 2 points or no = 0 points). The maximum disability score in this inventory is 100 points. The Spanish adaptation was performed by Rodríguez et al. in 2000, and provides a good index of internal consistency (Cronbach 0.94).

SECONDARY OUTCOMES:
Cervical range of motion | 8 weeks
  A cervical range of motion (CROM) device was used to assess range of motion of the cervical spine. Higher inter-tester reliability for the CROM is reported for measures of the upper cervical spine ICC> = 0.89. To assess upper cervical flexion and extension, the patient was standing with the back against the wall, looking forward horizontally and performed upper cervical flexion and extension guided by the examiner. For the assessment of cervical flexion and extension, the patient was seated and performed the movements whilst the examiner placed one hand on the sternum and the other over the upper thoracic region to minimise compensatory movements.

REFERENCES:
- [Background] Victoria Espi-Lopez G, Arnal-Gomez A, Arbos-Berenguer T, Gonzalez AAL, Vicente-Herrero T. Effectiveness of Physical Therapy in Patients with Tension-type Headache: Literature Review. J Jpn Phys Ther Assoc. 2014;17(1):31-38. doi: 10.1298/jjpta.Vol17_005. PMID 25792906
- [Background] Espi-Lopez GV, Gomez-Conesa A, Gomez AA, Martinez JB, Pascual-Vaca AO, Blanco CR. Treatment of tension-type headache with articulatory and suboccipital soft tissue therapy: A double-blind, randomized, placebo-controlled clinical trial. J Bodyw Mov Ther. 2014 Oct;18(4):576-85. doi: 10.1016/j.jbmt.2014.01.001. Epub 2014 Jan 10. PMID 25440210
- [Background] Espi-Lopez GV, Gomez-Conesa A. Efficacy of manual and manipulative therapy in the perception of pain and cervical motion in patients with tension-type headache: a randomized, controlled clinical trial. J Chiropr Med. 2014 Mar;13(1):4-13. doi: 10.1016/j.jcm.2014.01.004. PMID 24711779
- [Result] Espi-Lopez GV, Rodriguez-Blanco C, Oliva-Pascual-Vaca A, Benitez-Martinez JC, Lluch E, Falla D. Effect of manual therapy techniques on headache disability in patients with tension-type headache. Randomized controlled trial. Eur J Phys Rehabil Med. 2014 Dec;50(6):641-7. Epub 2014 Apr 30. PMID 24785463